CLINICAL TRIAL: NCT05119816
Title: Effect of Music Therapy Intervention on Heart Rate, Anxiety and Pain During Kidney Biopsy: a Randomized Controlled Trial.
Brief Title: Music Therapy Intervention During Kidney Biopsy.
Acronym: MTI-KB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Loreto Gesualdo, MD, professor, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0033297/06/05/2020
Record Dates: First submitted 2021-11-04; First posted 2021-11-15 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Kidney Diseases; Kidney Dysfunction; Kidney Disease, Chronic
Keywords: music therapy; anxiety; pain; heart rate variability; satisfation
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy group (Experimental): Patients receive an individual intervention of receptive music therapy during biopsy
  Interventions: Other: music therapy intervention
- Control group (No Intervention): Patients receive standard care

INTERVENTIONS:
Other: music therapy intervention — Received a customize playlists prepared by a certified music therapist to listening to during KB
  Arms: music therapy group

SUMMARY:
Kidney biopsy (KB) is an invasive procedure that is very useful in diagnosing kidney disease in both the native kidney and the transplanted kidney. Patients undergo KB can feel anxiety and pain. Pain is considered one of the worst experiences for patients and anxiety affects the sympathetic nervous system, the endocrine system and the immune system. The aim of this preliminary study was to evaluate the influence of MTI as a complementary/nonpharmacological intervention on heart rate variability, anxiety and pain and promote more compliant behaviours during KB.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* not severe neurological or psychiatric conditions
* not hearing impairment

Exclusion Criteria:

* age under 18 years
* severe neurological or psychiatric conditions
* hearing impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory Y-1 | 30 minutes before biopsy
  State Trait Anxiety Inventory Y-1(STAI-Y1) was used to measure how the subject felt in that moment. Subjects were asked to rate the intensity of their anxious feelings on 20 items on a four point scale: not at all, somewhat, moderately so, or very much so. STAI-Y values <40 defined absence of anxiety, between 40 and 50 mild anxiety, 51-60 moderate anxiety, and> 59 severe anxiety. T0 30 minutes before biopsy
State Trait Anxiety Inventory Y-1 | 1 hour after biopsy
  State Trait Anxiety Inventory Y-1(STAI-Y1) was used to measure how the subject felt in that moment. Subjects were asked to rate the intensity of their anxious feelings on 20 items on a four point scale: not at all, somewhat, moderately so, or very much so. STAI-Y values <40 defined absence of anxiety, between 40 and 50 mild anxiety, 51-60 moderate anxiety, and> 59 severe anxiety. T1 1 hour after biopsy
visual analogic scale (VAS) | through study completion - 5 minutes after biopsy
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.

SECONDARY OUTCOMES:
heart rate variability | during biopsy procedure
  Heart rate variability (HRV) is a non-invasive measure reflecting the variation over time of the period between consecutive heartbeats (RR intervals) and has been proved to be a reliable marker of the autonomic nervous system(ANS) activity.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUConsorziale Policlinico Di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No